CLINICAL TRIAL: NCT04023357
Title: Marginal Integrity and Clinical Evaluation of Polyetheretherketone (PEEK) Versus Lithium Disilicate (E-max) Endocrowns.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed mohamed osman Youssef, Internal resident faculty of oral & dental medicine Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: emax_peek
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital | interventions — polyetheretherketone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK (Experimental): PEEKs (polyetheretherketones) are presented as alternative materials to metal and glass ceramics,1 Their elastic modulus comparable to those of cortical bone and dentin so the polymer could exhibit good stress distribution. Also they have high fracture resistance, and low abrasion to the antagonist enamel.
  Yet clinical studies are needed to evaluate their clinical performance.
  Interventions: Other: PEEK
- Emax (Active Comparator): lithium disilicate glass-ceramic which is etchable and proved to have good success rate if used for Endocrowns
  Interventions: Other: Emax

INTERVENTIONS:
Other: PEEK — New polyetheretherketones material
  Other Names: BioHPP polyetheretherketones
  Arms: PEEK
Other: Emax — standard etchable glass ceramic used for Endocrowns
  Other Names: lithium disilicate glass ceramic
  Arms: Emax

SUMMARY:
Patients need Endocrowns for their teeth usually use Emax as an etchable ceramic. Yet they have disadvantages that may influence the outcome of the endocrowns, among which is the high stiffness and rigidity owing to the higher modulus of elasticity (67.2 GPa)( compared to natural dentin (18.6 GPa) which may affect the marginal adaptation.so a less rigid material is needed. PEEKs (polyetheretherketones) are presented as alternative materials to metal and glass ceramics, Their elastic modulus comparable to those of cortical bone and dentin so the polymer could exhibit good stress distribution. Also they have high fracture resistance, and low abrasion to the antagonist enamel.

.but the investigators have to know clinically it is performance , so the investigators are going to have Parallel groups in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to be:

* From 18-60 years old, and able to read and sign the informed consent document.
* Physically and psychologically able to tolerate conventional restorative procedures
* Have no active periodontal or pulpal diseases.
* Willing to return for follow-up examinations and evaluation

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth
* Patient with fractured teeth of more than 50% enamel loss
* Patients with poor oral hygiene and motivation
* Pregnant women
* Psychiatric problems or unrealistic expectations
* Lack of opposite occluding dentition in the area intended for restoration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
evaluation of marginal gap | through study completion, an average of 1 year
  Marginal gap of the restorations assessed by Silicon replica technique using digital microscope

SECONDARY OUTCOMES:
Clinical evaluation of marginal adaptation | 1 Year
  Marginal adaptation of the restorations assessed clinically using dental mirror and probe according to the modified united states public health service criteria (USPHS)
Clinical evaluation of fracture resistance | 1 Year
  Fracture resistance of the restorations assessed clinically using dental mirror and probe according to the modified united states public health service criteria (USPHS)

OTHER OUTCOMES:
Clinical evaluation of Retention | 1 Year
  Retention of the restorations assessed clinically using dental mirror and probe according to the modified united states public health service criteria (USPHS)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Otto T, Mormann WH. Clinical performance of chairside CAD/CAM feldspathic ceramic posterior shoulder crowns and endocrowns up to 12 years. Int J Comput Dent. 2015;18(2):147-61. English, German. PMID 26110927
- [Background] Zoidis P, Bakiri E, Polyzois G. Using modified polyetheretherketone (PEEK) as an alternative material for endocrown restorations: A short-term clinical report. J Prosthet Dent. 2017 Mar;117(3):335-339. doi: 10.1016/j.prosdent.2016.08.009. Epub 2016 Sep 28. PMID 27692583
- [Background] Sevimli G, Cengiz S, Oruc MS. Endocrowns: review. J Istanb Univ Fac Dent. 2015 Apr 29;49(2):57-63. doi: 10.17096/jiufd.71363. eCollection 2015. PMID 28955538